CLINICAL TRIAL: NCT07200947
Title: A Phase II Clinical Trial of Iparomlimab and Tuvonralimab in Combination With Platinum-based Chemotherapy in Patients With SMARCA4-Deficient, Locally Advanced or Metastatic Non-Small Cell Lung Cancer.
Brief Title: A Phase II Study of QL1706 and Platinum-Based Chemotherapy in Patients With SMARCA4-Deficient, Locally Advanced or Metastatic Non-Small Cell Lung Cancer.
Acronym: QL1706
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhijie Wang (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor-Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5684
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: SMARCA4-Deficient Tumor; Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: QL1706; combination therapy; first line therapy; SMARCA4-Deficient Locally advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): This study evaluates a first-line treatment for locally advanced or metastatic SMARCA4-deficient non-small cell lung cancer (NSCLC), combining QL1706-a bifunctional antibody targeting both PD-1 and CTLA-4-with platinum-based chemotherapy (nab-paclitaxel + carboplatin). QL1706 is designed to provide dual immune checkpoint blockade with a optimized safety profile. This synergistic approach integrates immunotherapy and chemotherapy to address the high unmet need in this aggressive disease subset. Patients receive QL1706 monotherapy as maintenance treatment after 4-6 cycles of induction. No prior prospective studies have evaluated this regimen in SMARCA4-deficient NSCLC.
  Interventions: Drug: QL1706, nab-paclitaxel, carboplatin

INTERVENTIONS:
Drug: QL1706, nab-paclitaxel, carboplatin — Participants will receive QL1706 (5 mg/kg, IV, day 1) in combination with nab-paclitaxel (260 mg/m², IV, day 1) and carboplatin (AUC=4-5, IV, day 1) every 21 days for 4-6 cycles. Dose adjustments may be made based on clinical judgment. Patients who do not experience disease progression or intolerable toxicity will proceed to maintenance therapy with QL1706 (5 mg/kg, IV, day 1) every 21 days. Treatment will continue until disease progression, unacceptable toxicity, consent withdrawal, investigator decision, loss to follow-up, death, or meeting other protocol-defined criteria for discontinuation. The maximum duration of QL1706 treatment is 24 months, after which continuation will be at the investigator's discretion based on individual benefit-risk assessment.

SUMMARY:
This single-arm, open-label, Phase II study assesses first-line QL1706 (iparomlimab and tuvonralimab, an anti-PD-1/CTLA-4 bispecific antibody) combined with platinum-based chemotherapy to treat patients with treatment-naïve, locally advanced or metastatic, SMARCA4-deficient non-small cell lung cancer (NSCLC).

The main questions it aims to answer are:Evaluate the efficacy and safety of this combination regimen in this specific patient population. Explore correlations between tumor molecular characteristics, the immune microenvironment, and treatment efficacy or toxicity.

Participants must:

Have histologically or cytologically confirmed, treatment-naïve, locally advanced or metastatic non-small cell lung cancer (NSCLC) with SMARCA4 deficiency. Be willing to provide archived or fresh tumor tissue samples. If unavailable, enrollment may proceed per investigator assessment. Have at least one measurable lesion per RECIST v1.1.

DETAILED DESCRIPTION:
SMARCA4-deficient non-small cell lung cancer (NSCLC) represents a highly aggressive molecular subtype, accounting for approximately 5-10% of all NSCLC cases. The majority of patients (over 80%) present with distant metastases at diagnosis, and prognosis is exceptionally poor, with median overall survival (mOS) historically ranging from 4 to 7 months. Currently, no standardized treatment exists for this subset, and therapeutic efficacy remains limited.

Immune checkpoint inhibitors (ICIs) combined with platinum-based chemotherapy have become a cornerstone of treatment for advanced NSCLC without driver mutations. However, the benefit of this approach in SMARCA4-deficient NSCLC is uncertain and appears heterogeneous. A large retrospective analysis (n=707) indicated that SMARCA4-mutant tumors derived significantly less benefit from first-line chemoimmunotherapy compared to wild-type tumors, showing inferior objective response rate (ORR) and progression-free survival (PFS). Conversely, other retrospective data suggest a potential survival advantage with ICI-chemotherapy over chemotherapy alone. This discrepancy may be influenced by BRG1 protein expression loss, a key molecular feature with prognostic implications, highlighting the complexity of this disease and the need for prospective validation.

QL1706 (iparomlimab and tuvonralimab) is a novel bifunctional MabPair antibody that concurrently targets PD-1 and CTLA-4 at a fixed 2:1 ratio. This design aims to enhance synergistic immune activation while potentially mitigating toxicity associated with conventional CTLA-4 inhibition. Approved in 2024, QL1706 has demonstrated promising efficacy and a manageable safety profile in multiple solid tumors, including NSCLC. In the DUBHE-L-201 trial, QL1706 combined with chemotherapy demonstrated encouraging activity.

To date, there are no prospective clinical data on the use of QL1706 combined with chemotherapy in SMARCA4-deficient NSCLC. This phase II, single-arm, open-label trial is proposed to evaluate the efficacy and safety of QL1706 plus platinum-based chemotherapy as a first-line treatment for patients with locally advanced or metastatic SMARCA4-deficient NSCLC. The study aims to address a significant unmet need and explore a potentially effective therapeutic strategy for this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

1. Voluntary participation and provision of signed written informed consent.
2. Age ≥ 18 years.
3. Life expectancy ≥ 3 months.
4. Histologically or cytologically confirmed diagnosis of Stage IIIB-IV lung cancer that is not amenable to curative surgery or radiotherapy.
5. Tumor demonstrates loss of BRG1 protein (encoded by the SMARCA4 gene) as confirmed by immunohistochemistry (IHC).
6. No prior systemic anti-cancer therapy for advanced disease.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Willingness to provide archived or fresh tumor tissue samples from primary or metastatic lesions. If unavailable, enrollment may be permitted following investigator assessment.
9. At least one measurable lesion as defined by RECIST v1.1.
10. Adequate organ function within the screening period, as evidenced by:

10.1 Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L 10.2 Platelet count ≥ 100 × 10^9/L 10.3 Hemoglobin ≥ 90 g/L (without transfusion within 14 days) 10.4 Serum creatinine ≤ 1 × ULN OR Creatinine clearance > 50 mL/min (calculated by Cockcroft-Gault formula) 10.5 AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastases) 10.6 Total bilirubin ≤ 1.5 × ULN (except for participants with Gilbert's syndrome) 10.7 TSH, FT3, and FT4 within normal limits (±10%)

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Pathological diagnosis containing a small cell component.
2. Symptomatic brain metastases.
3. Leptomeningeal metastases.
4. Recurrence within 6 months after completing prior adjuvant therapy (if applicable).
5. Active, known, or suspected autoimmune disease (with specific exceptions, e.g., vitiligo, type I diabetes, hypothyroidism managed with hormone replacement only).
6. Active tuberculosis (TB) infection or history of active TB within the past year.
7. Comorbidities requiring immunosuppressive medications, including systemic corticosteroids at immunosuppressive doses.
8. Pregnancy or lactation in female participants.
9. Symptomatic interstitial lung disease that could interfere with the detection or management of suspected drug-related pulmonary toxicity.
10. Known HIV infection, active Hepatitis B (HBsAg positive with HBV-DNA > 10^3 copies/mL), or active Hepatitis C (HCV antibody positive with detectable HCV-RNA).
11. Significant history of neurological or psychiatric disorders.
12. Treatment with any investigational drug within 4 weeks prior to the first dose of study treatment.
13. Use of Chinese herbal medicines with anti-tumor activity within 2 weeks prior to study treatment initiation.
14. History of another active malignancy within the past 2 years (with specific exceptions for certain early-stage cancers).
15. Significant cardiovascular or cerebrovascular disease history.
16. Uncontrolled thrombotic events within 6 months prior to screening.
17. Administration of a live vaccine within 28 days prior to the first study dose.
18. Major surgery or significant trauma within 4 weeks prior to the first study dose.
19. Conditions that may impair oral drug absorption.
20. Uncontrolled active infection requiring systemic therapy.
21. Known hypersensitivity to any of the study drug components.
22. Any other condition that, in the investigator's judgment, would make the participant unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the end of monitoring at 2 years.
  PFS is defined as the time from the first dose of study treatment to the first documentation of disease progression according to RECIST v1.1 (as assessed by investigators) or death from any cause, whichever occurs first. Subjects who are alive without progression at the time of analysis will be censored at the date of the last tumor assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of monitoring at 2 years.
  OS is defined as the time from the first dose of study treatment to death from any cause. Subjects who are alive at the time of analysis will be censored at the date of last follow-up.
Objective Response Rate (ORR) | From enrollment to the end of monitoring at 2 years.
  ORR is defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR) as per RECIST v1.1.
Duration of Response (DoR) | From enrollment to the end of monitoring at 2 years.
  DoR is defined as the time from the first documentation of CR or PR to the first documentation of disease progression or death.
Disease Control Rate (DCR) | From enrollment to the end of monitoring at 2 years.
  DCR is defined as the proportion of subjects who achieve CR, PR, or stable disease (SD) as their best overall response.
The incidence of adverse events | From enrollment to the end of monitoring at 2 years
  Incidence, nature, and severity of adverse events (AEs), graded according to NCI-CTCAE v5.0, including immune-related AEs and serious AEs.

OTHER OUTCOMES:
Immune-Related Adverse Events (irAEs) | From enrollment to the end of monitoring at 2 years
  Occurrence and grade of immune-related adverse events as defined by pre-specified criteria, including rash, colitis, hepatitis, endocrinopathies, and pneumonitis.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No